CLINICAL TRIAL: NCT04908007
Title: Institutional Management and Professional Experience During the Pandemic COVID-19 by Health Care Institutions in the Auvergne-Rhône-Alpes Region: Assessment and Lessons Learned
Brief Title: COvid Pandemic Institutional maNaGement
Acronym: COPING
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0466
Record Dates: First submitted 2021-05-17; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-04

CONDITIONS: Covid19
Keywords: Covid-19; Institutional management process; Professional experience; Crisis management
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Professional qualitative group: Qualitative analysis of crisis management by interviewing professionals most involved during the crisis in each university hospital.
  Interventions: Other: Qualitative analysis for professionals
- Professional quantitative group: Quantitative analysis of crisis management using the WHO grid adapted sent to the target persons identified within the establishments
  Interventions: Other: Quantitative analysis for Professionals
- Patient quantitative group: Quantitative analysis of crisis management using a questionnaire sent to patients hospitalized in the first wave asking them about their perception of crisis and post-crisis management.
  Interventions: Other: Quantitative analysis for Patients
- Tools development: Development of tools to prepare for situations of uncertainty
  Interventions: Other: Tools development

INTERVENTIONS:
Other: Qualitative analysis for professionals — 3 individual interviews with the different categories of professionals most involved during the crisis in each university hospital. In the first phase, the points of improvement identified will be analyzed In the second phase, good practices and innovations will be analyzed. For these first two phases, the duration of one hour was chosen because it is difficult to mobilize the professionals for longer. Individual interviews are preferred, but group interviews are possible with no more than three people so that everyone can express himself or herself. Finally, individual interviews of 15 to 30 minutes will be conducted with some of the people interviewed previously in order to identify the costs of the dysfunctions or problems encountered during the crisis.
  Questionnaires with establishments associated with the crisis management, the ARS AuRA and France Assos Santé AuRA.
  Analysis of evidence documents in the university hospitals
  Groups: Professional qualitative group
Other: Quantitative analysis for Professionals — A self-assessment of the three phases of the crisis management process (preparation, crisis management, crisis recovery) will be carried out in the participating establishments using the WHO grid with the target persons identified within the establishments.
  This step will use the crisis response assessment tool developed by the WHO following the H1N1 pandemic in 2011. This grid will be adapted beforehand to the COVID-19 situation and to the local organization by the study's scientific committee. The dimensions investigated will be : Command and control, Communication, Safety and security, Triage, Surge capacity, Continuity of essential services; Human resources, Logistics and supply management, Post-disaster recovery.
  The grids will be sent to the 4 university hospitals to be filled in with the target audience recommended by the WHO methodological guide.
  The results of this self-assessment will be linked to and interpreted with the results of the interviews in phase 1.
  Groups: Professional quantitative group
Other: Quantitative analysis for Patients — A questionnaire of patients' perceptions on the same perimeter (crisis and post-crisis management, from the point of view of points of improvement and good practices) will be constructed and sent by the management of the establishments to all patients hospitalized for 48 hours or more during the first wave and who have left their email address (methods similar to the e-satis survey). The online questionnaire survey is preferred in order to get away from the emotion and for feasibility reasons. This patient experience questionnaire adapted to COVID will be co-constructed with expert/partner patients and user associations.
  Four dimensions will be investigated : The perception of the quality of the information received by the patient, The nature of the information on the specific health protection protocol from which the patient benefited, The patient's consideration of the overall context, during and after, The effects of the health context on the overall management of the patient
  Groups: Patient quantitative group
Other: Tools development — Development of tools to prepare for situations of uncertainty : In the third phase of the project, design thinking workshops will be organized (within the HCL) to develop training (in the form of simulation) in order to appropriate virtuous practices in situations of uncertainty. The purpose of these training sessions will be to improve the institution's ability to learn in a situation of uncertainty and thus to develop its reliability.
  The aim of these workshops is to provide tools for raising awareness of situations of uncertainty to all hospital staff.
  Groups: Tools development

SUMMARY:
Covid-19 has increased organizational tensions within health services (lack of resources, difficulties in recruiting healthcare professionals , elderly and polypathological patients, etc.) and tested the reliability of health facilities. This project aims to draw lessons so that hospitals can transform themselves while improving their reliability to face future crises and other exceptional situations.

Research hypothesis:

Crisis management arrangements lack sensitivity to uncertainty, which manifests itself in lower quality of care and efficiency losses for the entire institution.

The virtuous practices implemented during the crisis spontaneously incorporated principles of the highly reliable organization.

The integration of principles from complexity theory into the management of institutions promotes high reliability organization.

Sustaining these virtuous practices in order to anticipate and cope with crises requires the activation of two interconnected levers: a shared vision (by patients, healthcare professionals, ARS, HAS, and the Ministry in the first place) of the meaning of the action taken by hospitals, and the development of a policy enabling hospitals to become both learning and highly reliable.

Main objective:

To evaluate the management process of the Covid-19 epidemic by the university hospitals of the Auvergne-Rhône-Alpes region, and the structures linked to them (establishments in their territory, ARS, user associations), in terms of points of improvement and good practices. This evaluation concerns the preparation, management and exit phases of the crisis.

ELIGIBILITY:
Inclusion Criteria:

* Establishments :

  * 4 university hospitals: Lyon, St Etienne, Clermont Ferrand, Grenoble
  * Establishments in the same territories, public and private
* Professionals and members of the institutions' bodies:

  * Governance: management and chair of the CME
  * Management (care, communication, medical, technical, logistics, IT, personnel)
  * Clinical and public health cluster governance
  * Medical, paramedical and non-medical staff in the departments most concerned (emergency and EMS reception, intensive care, infectiology, hygiene, virology, imaging, occupational medicine in particular)
  * Organizations representing the personnel
  * Members of the users' representatives committee
* Adult patients hospitalized for at least 48 hours during the study period (quantitative study by questionnaires).

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Professionals and members of the institutions' bodies in the 4 university hospitals: Lyon, St Etienne, Clermont Ferrand, Grenoble
  * Adult patients hospitalized for at least 48 hours during the first wave of the pandemic COVID-19 in the 4 university hospitals: Lyon, St Etienne, Clermont Ferrand, Grenoble
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Crisis management process based on a qualitative approach | The Qualitative analysis (intervention 1) will take place from September, 2020 to December, 2021
  The qualitative evaluation (interviews, document review) will make it possible to identify the points of improvement and virtuous practices implemented in the establishments.
Crisis management process based on a quantitative approach with the professionals (identified within the establishments) | The Quantitative analysis for professionals (intervention 2) will be conducted from March, 2021 to June 2021.
  The quantitative evaluation will be based on the WHO checklist. This first part will report, for each hospital, the proportion of items validated in each dimension of the WHO checklist (https://www.who.int/publications/i/item/hospital-emergency-response-checklist):
Crisis management process based on a quantitative approach with the patients (hospitalized in the first wave) | The Quantitative analysis for patients (intervention 3) will be conducted from March, 2021 to June 2021. The tool development phase (intervention 4) will be carried out from January, 2022 to June, 2022
  The second quantitative evaluation will be based on patients' perceptions with a constructed questionnaire on theses perimeters: crisis and post-crisis management, from the point of view of points of improvement and good practices.
  This patient experience questionnaire will be adapted to COVID with expert/partner patients and user associations.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU Clermont-Ferrand , Pôle de Santé Publique, unité d'Epidémiologie, Economie de la Santé et Prévention, Clermont-Ferrand
  - CHU Grenoble, Pôle Santé Publique, service de veille sanitaire, Grenoble
  - Hospices Civils de Lyon, DOQ-RU, Lyon
  - CHU Saint-Etienne , Unité de gestion du risque infectieux, Saint-Etienne